CLINICAL TRIAL: NCT04165928
Title: Multicenter Study of Tetanus Patients in Fujian Province of China
Status: Completed | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xiuling Shang, Deputy Director of the Physician, Fujian Provincial Hospital
Other Study IDs: K2018-09-005
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Tetanus
Keywords: neonatal tetanus; tetanus immunization program; drug-induced; tetanus antitoxin; critical care medicine; artificial airway
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Tetanus is a life-threatening disease in developing countries, and accompanied by a high mortality rate. China is the world's largest developing country, and Fujian Province is a typical coastal province in China with a relatively developed economy. Therefore, the purpose of this study was to investigate the epidemiology, incidence and management of tetanus in Fujian Province and to understand the current treatment and prognosis of tetanus patients in China.

Methods: This was a retrospective multicenter observational study of patients who presented with a clinical diagnosis of tetanus at 5 general hospitals in Fujian. Data was analyzed using computer software system.

ELIGIBILITY:
Inclusion Criteria:

* This study included all patients of all age groups and both sexes who presented with a clinical diagnosis of tetanus.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included all patients of all age groups and both sexes who presented with a clinical diagnosis of tetanus.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Outcomes of the tetanus patients | 2008-01-01~2018-10-31
  The survival data of tetanus patients.

SECONDARY OUTCOMES:
The hospitalization time. | 2008-01-01~2018-10-31
  The total length of hospitalization and the length of stay in the ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China